CLINICAL TRIAL: NCT01090141
Title: Pharmacokinetic Analysis of Micafungin in Overweight, Obese, and Extremely Obese Volunteers
Brief Title: Drug Concentration Analysis of Micafungin in Overweight, Obese, and Extremely Obese Volunteers
Acronym: Micafungin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJ-07-003
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Nutrition Disorders; Overweight
Keywords: Micafungin; Body Weight; Anti-Infective Agents; Signs and Symptoms; Mycoses; Therapeutic Uses; Antifungal Agents; Overnutrition; Pharmacologic Actions
MeSH Terms: conditions — Obesity; Nutrition Disorders; Overweight; Body Weight; Signs and Symptoms; Mycoses; Overnutrition | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subjects recieving 100 mg of Micafungin (Active Comparator)
  Interventions: Drug: Micafungin
- Subjects recieving 300 mg of Micafungin (Active Comparator)
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — 100 mg IV infusion over 1 hour
  Arms: Subjects recieving 100 mg of Micafungin
Drug: Micafungin — 300 mg IV infusion over 1 hour
  Arms: Subjects recieving 300 mg of Micafungin

SUMMARY:
The purpose of this study is to assess the drug concentration of Micafungin amongst healthy volunteers having different weight groups.

DETAILED DESCRIPTION:
This is a single center study. A total of 36 adult volunteers will be consented for the study. Volunteers will be admitted for an overnight stay. Half will be female and half male. Twelve volunteers will have a body mass index (BMI) less than 25 kg/m2, 12 will have a BMI 25-40 kg/m2, and 12 will have a BMI greater than 40 kg/m2. Volunteers will have height and weight measured after they have consented to participate. Exactly half the volunteers in each category will received a single dose of intravenous micafungin of 100 mg, while the other half will receive 300 mg as determined by a coin flip. The volunteers will have blood drawn via an intravenous catheter just prior to the dose, and then at 1, 4, 8, 12, 16, and 24h after the drug dose. The intravenous catheter is then removed after the 24h blood draw, and the volunteer discharged from the study. Compensation will be provided to the participants for their time.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* 18 years or older
* All racial and ethnic origins
* English or Spanish speaking

Exclusion Criteria:

* Pregnant or nursing or unwilling to use a reliable contraception method during the study. The effects of micafungin on pregnancy are unknown. In addition, the metabolic changes that accompany pregnancy may alter the concentration-time profile of micafungin, so that the pregnancy and post-partum state would be a confounding variable.

  * Abnormal liver function tests: transaminases>10 times upper limit of normal, Alkaline phosphatase>5 times upper limit of normal, total bilirubin>5 times upper limit of normal.
* Creatinine Clearance < 70 ml/min as estimated by the Cockcroft-Gault equation
* History of allergies to echinocandins
* Echinocandins are contraindicated for any reason
* Volunteers unwilling to comply with study procedures.
* Suspected or documented systemic fungal infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tawanda Gumbo, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI (Tawanda Gumb) has left the institution. Since May 2020, we tried to locate original PI and reached out to two PRS administrators at Baylor, Texas Tech University where we believe the original PI is, but they have informed us PI is no longer there, and they do not know where data are for this study. Further efforts were made to locate manuscript, and study team members, but were unsuccessful. No study data are available
Period: Overall Study
Arm/Group | Subjects Recieving 100 mg of Micafungin | Subjects Recieving 300 mg of Micafungin
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI (Tawanda Gumb) has left the institution. Since May 2020, we tried to locate original PI and reached out to two PRS administrators at Baylor, Texas Tech University where we believe the original PI is, but they have informed us PI is no longer there, and they do not know where data are for this study. Further efforts were made to locate manuscript, and study team members, but were unsuccessful. No study data are available
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Recieving 100 mg of Micafungin | Subjects Recieving 300 mg of Micafungin | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Serum Clearance of Micafungin
Time Frame: 0-24 Hrs
Population: as for baseline characteristics
Arm/Group | Subjects Recieving 100 mg of Micafungin | Subjects Recieving 300 mg of Micafungin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The PI (Tawanda Gumb) has left the institution.Since May 2020, we tried to locate original PI and reached out to two PRS administrators at Baylor, Texas Tech University where we believe the original PI is, but they have informed us PI is no longer there, and they do not know where data are for this study. Further efforts were made to locate manuscript, and study team members, but were unsuccessful. No study data are available
Arm/Group | Subjects Recieving 100 mg of Micafungin | Subjects Recieving 300 mg of Micafungin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The PI (Tawanda Gumb) has left the institution. Since May 2020, we tried to locate original PI and reached out to two PRS administrators at Baylor, Texas Tech University where we believe the original PI is, but they have informed us PI is no longer there, and they do not know where data are for this study. Further efforts were made to locate manuscript, and study team members, but were unsuccessful. No study data are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No